CLINICAL TRIAL: NCT01373216
Title: EXEnatide in Patients Undergoing Coronary Artery Bypass Grafting for Improved glUcose conTrol and hemodynamIc ValuEs
Brief Title: Glucagon-like Peptide 1 Agonist Exenatide for Improved Glucose Control and Cardiac Function in Patients With Aortocoronary Bypass
Acronym: Executive
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Martin Haluzik, Prof. Martin Haluzik, MD DSc, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H8O-CY-O027
Record Dates: First submitted 2011-06-10; First posted 2011-06-14 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Coronary Artery Disease; Decreased Left Ventricular Function
MeSH Terms: conditions — Coronary Artery Disease; Ventricular Dysfunction, Left | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exenatide (Experimental): Patients with decreased left ventricular function undergoing elective coronary artery by-pass grafting receiving perioperatively i.v. exenatide on top of standard treatment
  Interventions: Drug: Exenatide
- Control (No Intervention): Patients with decreased left ventricular function undergoing elective coronary artery by-pass grafting receiving standard treatment

INTERVENTIONS:
Drug: Exenatide — Perioperative continuous i.v. administration of exenatide lasting for 72 hours - 40 ng/min for initial 30 min, 20 ng/min for remaining 71.5 hours
  Arms: Exenatide

SUMMARY:
GLP-1 has not only beneficial effects on glucose metabolism but also direct positive effects on cardiac function and metabolism in both experimental models and in patients with type 2 diabetes mellitus. Clinical data on the effects of GLP-1 agonists on cardiac function and glucose control in patients undergoing cardiac surgery are not known. Based on the results of experimental studies there is a potential for exenatide to positively influence both cardiac function and glucose metabolism in cardiac surgery patients with and without type 2 diabetes mellitus. The primary endpoint of this study is to examine whether pre- and peri-operative administration of exenatide affects perioperative hemodynamics, echocardiographic parameters, necessity of antiarrhythmic and inotropic treatment and glucose control in patients with coronary atherosclerosis and decreased left ventricular function undergoing elective coronary artery bypass grafting operation (CABG). In addition, safety and tolerability of peri-operative administration of exenatide in these patients will be examined as a secondary study objective.

ELIGIBILITY:
Inclusion Criteria:

* elective coronary artery bypass grafting operation (CABG)
* decreased left ventricular (LV) systolic function (EF LV ≤ 50%)
* Age 18 to 85
* Signed informed consent
* Females with childbearing potential have to use appropriate contraceptive measures during the whole study period and 6 months after terminating exenatide infusion (hormonal contraception or double-barrier contraception for both partners)

Exclusion Criteria:

* allergy to exenatide
* allergy to insulin
* mental incapacity or language barrier
* use of incretin-based therapies <3 months before inclusion in the study
* diabetic ketoacidosis
* established autonomic neuropathy
* history of acute pancreatitis or severe disease of digestive tract
* renal failure (preoperative creatinine ≥ 180 umol/l)
* liver failure (coagulation times more than 1.5 times higher without use of anticoagulants)
* cardiac surgical procedure on valve, thoracic aorta or MAZE procedure
* pregnancy and lactation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-06; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Cardiac function - echocardiographic parameters | 90 days after administration of exenatide
  * cardiac chamber dimensions
  * left ventricular systolic function
  * left ventricular diastolic function
  * right ventricular systolic function

SECONDARY OUTCOMES:
Number of participants with adverse effects | 90 days after administration of exenatide

CONTACTS AND LOCATIONS:
Overall Officials: Martin Haluzik, D.Sc., Principal Investigator — General University Hospital, Charles University, Prague
Locations (1):
- General University Hospital, Prague, Czechia

REFERENCES:
- [Derived] Lips M, Mraz M, Klouckova J, Kopecky P, Dobias M, Krizova J, Lindner J, Diamant M, Haluzik M. Effect of continuous exenatide infusion on cardiac function and peri-operative glucose control in patients undergoing cardiac surgery: A single-blind, randomized controlled trial. Diabetes Obes Metab. 2017 Dec;19(12):1818-1822. doi: 10.1111/dom.13029. Epub 2017 Jul 31. PMID 28581209